CLINICAL TRIAL: NCT06242392
Title: The Correlation Between Homologous Recombination Deficiency Detection and the Efficacy of PARP Inhibitors in Ovarian Cancer
Brief Title: The Correlation Between HRD Detection and the Efficacy of PARP Inhibitors in Ovarian Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Fujian Cancer Hospital (Other Government)
Collaborators: Fujian Provincial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ChenJian2
Record Dates: First submitted 2024-01-29; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Neoplasms
Keywords: Ovarian Neoplasms; homologous recombination deficiency; prognosis; Cost-effectiveness analysis
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- effective group: The tumor size of each diameter of the tumor before and after treatment was measured on magnetic resonance imaging or CT. According to Recist 1.1 criteria, patients who were evaluated as complete remission, partial remission and stable disease were included in the effective group. Patients assessed as having progressive disease were included in the treatment-refractory group.
  Interventions: Genetic: homologous recombination deficiency
- ineffective group: The tumor size of each diameter of the tumor before and after treatment was measured on magnetic resonance imaging or CT. According to Recist 1.1 criteria. Patients assessed as having progressive disease were included in the ineffective group.
  Interventions: Genetic: homologous recombination deficiency

INTERVENTIONS:
Genetic: homologous recombination deficiency — Homologous Recombination Deficiency (HRD) refers to a disruption or deficiency in the homologous recombination repair (HRR) pathway, which is a crucial mechanism in cells for repairing DNA double-strand breaks (DSBs). This pathway is particularly important for maintaining genomic stability.

SUMMARY:
Clinicopathological data were collected from ovarian cancer patients treated with PARP inhibitors, with follow-up imaging conducted before and after treatment. The efficacy was evaluated according to RECIST criteria, comparing the correlation between different HRD statuses and the efficacy of PARP inhibitors in ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ovarian cancer (any histological type) and possessing complete pathological hematoxylin and eosin (HE) stained slides and paraffin-embedded tissue blocks.
* Patients must be 18 years of age or older.
* Patients should not have concurrent multiple primary cancers.
* Patients must undergo an MRI or CT scan prior to starting treatment.
* According to RECIST (Response Evaluation Criteria In Solid Tumors) criteria, patients must have at least one measurable lesion.
* Participants must provide informed consent, voluntarily cooperate with clinical follow-up, and sign an informed consent form.

Exclusion Criteria:

* Patients who do not have accessible tumor tissue required for Homologous Recombination Deficiency (HRD) testing.
* Patients whose clinical records are incomplete, making it impossible to effectively compare treatment efficacy.
* Patients who are lost to follow-up and for whom subsequent treatment outcomes cannot be tracked.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Ovarian Cancer who were treated from June 2020 to December 2026 and met the above inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-01-31 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of PARP inhibitors in the treatment of ovarian cancer | 2026-5-1
  Progression-Free Survival (PFS) is used to evaluate the efficacy of PARP inhibitor treatment in ovarian cancer with different HRD (Homologous Recombination Deficiency) statuses.

SECONDARY OUTCOMES:
cost-effectiveness analysis of using PARP inhibitors to treat cervical cancer | 2026-5-1
  The main economic outcome is the ICER.Health benefits were expressed as life years (LYs), and quality-adjusted life-years (QALYs) gained. The ICER was calculated by dividing the incremental cost difference between the two strategies, by the incremental difference in health outcomes (LYs and QALYs). Probabilistic Sensitivity Analysis (PSA) was performed to assess the impact of uncertainty around the key parameters of the model on the ICER. A second-order Monte Carlo simulation with 1000 iterations was used to run replicated outcomes. The normal distributions used for costs, utility and reimbursement ratio were carried to the specific limits.
PARP inhibitors in the treatment of ovarian cancer | 2026-5-1
  Overall survival (OS) was used toevaluate the efficacy of PARP inhibitor treatment in ovarian cancer with different HRD (Homologous Recombination Deficiency) statuses.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller RE, Leary A, Scott CL, Serra V, Lord CJ, Bowtell D, Chang DK, Garsed DW, Jonkers J, Ledermann JA, Nik-Zainal S, Ray-Coquard I, Shah SP, Matias-Guiu X, Swisher EM, Yates LR. ESMO recommendations on predictive biomarker testing for homologous recombination deficiency and PARP inhibitor benefit in ovarian cancer. Ann Oncol. 2020 Dec;31(12):1606-1622. doi: 10.1016/j.annonc.2020.08.2102. Epub 2020 Sep 28. PMID 33004253
- [Background] Vergote I, Gonzalez-Martin A, Ray-Coquard I, Harter P, Colombo N, Pujol P, Lorusso D, Mirza MR, Brasiuniene B, Madry R, Brenton JD, Ausems MGEM, Buttner R, Lambrechts D; European experts' consensus group. European experts consensus: BRCA/homologous recombination deficiency testing in first-line ovarian cancer. Ann Oncol. 2022 Mar;33(3):276-287. doi: 10.1016/j.annonc.2021.11.013. Epub 2021 Dec 1. PMID 34861371
- [Background] Lheureux S, Gourley C, Vergote I, Oza AM. Epithelial ovarian cancer. Lancet. 2019 Mar 23;393(10177):1240-1253. doi: 10.1016/S0140-6736(18)32552-2. PMID 30910306
- [Background] Doig KD, Fellowes AP, Fox SB. Homologous Recombination Repair Deficiency: An Overview for Pathologists. Mod Pathol. 2023 Mar;36(3):100049. doi: 10.1016/j.modpat.2022.100049. Epub 2023 Jan 10. PMID 36788098
- [Background] Ray-Coquard I, Pautier P, Pignata S, Perol D, Gonzalez-Martin A, Berger R, Fujiwara K, Vergote I, Colombo N, Maenpaa J, Selle F, Sehouli J, Lorusso D, Guerra Alia EM, Reinthaller A, Nagao S, Lefeuvre-Plesse C, Canzler U, Scambia G, Lortholary A, Marme F, Combe P, de Gregorio N, Rodrigues M, Buderath P, Dubot C, Burges A, You B, Pujade-Lauraine E, Harter P; PAOLA-1 Investigators. Olaparib plus Bevacizumab as First-Line Maintenance in Ovarian Cancer. N Engl J Med. 2019 Dec 19;381(25):2416-2428. doi: 10.1056/NEJMoa1911361. PMID 31851799
- [Background] Moore KN, du Bois A. Homologous recombination deficiency testing in first-line ovarian cancer. Ann Oncol. 2022 Mar;33(3):231-233. doi: 10.1016/j.annonc.2021.12.013. Epub 2022 Jan 8. No abstract available. PMID 35017033